CLINICAL TRIAL: NCT05772208
Title: A Multicenter, Randomized Controlled Phase III Trial of Induction Plus Concurrent Chemoradiotherapy Plus Camrelizumab or Nimotuzumab Versus Induction Plus Concurrent Chemoradiotherapy in Locally Advanced Nasopharyngeal Carcinoma With Detectable EBV DNA After One Cycle GP Regime Neoadjuvant Chemotherapy
Brief Title: Intensified Treatments for Patients With Locally Advanced Nasopharyngeal Carcinoma With Detectable EBV DNA After One Cycle GP Regime Neoadjuvant Chemotherapy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Chaosu Hu, MD and PhD, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2110244-20
Record Dates: First submitted 2023-03-06; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: EBV DNA; camrelizumab; nimotuzumab
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — camrelizumab; nimotuzumab; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- the combination of camrelizumab and standard treatment (Experimental): camrelizumab 200mg q3w 2 cycle combinted with the second and third cycle neoajuvant chemotherapy and camrelizumab 200mg q3w 8 cycle starting one month after concurrent chemo-radiotherapy.
  Interventions: Drug: Camrelizumab; Drug: neoadjuvant chemotherapy and CCRT
- the combination of nimotuzumab and standard treatment (Experimental): nimotuzumab 200mg qw combined with the second and third cycle neoajuvant chemotherapy and nimotuzumab 200mg qw used during chemo-radiotherapy.
  Interventions: Drug: Nimotuzumab; Drug: neoadjuvant chemotherapy and CCRT
- standard treatment (Active Comparator): the second and third neoajuvant chemotherapy with GP regimen (gemcitabine 1g/m2 d1，8 plus cisplatin 75mg/m2 ) concurrent chemotherapy: single cisplatin (80mg/m2) for two cycle definitive radiotherapy for primay lesion and lymph node region.
  Interventions: Drug: neoadjuvant chemotherapy and CCRT

INTERVENTIONS:
Drug: Camrelizumab — camrelizumab 200mg q3w
  Arms: the combination of camrelizumab and standard treatment
Drug: Nimotuzumab — nimotuzumab 200mg qw
  Arms: the combination of nimotuzumab and standard treatment
Drug: neoadjuvant chemotherapy and CCRT — the second and third neoajuvant chemotherapy with GP regimen (gemcitabine 1g/m2 d1，8 plus cisplatin 75mg/m2 ) concurrent chemotherapy: single cisplatin (80mg/m2) for two cycle definitive radiotherapy for primay lesion and lymph node region.

SUMMARY:
The goal of this multicenter randomized non-inferior study is to compare the additon of camrelizumab or nimotuzumab to neoadjuvant chemotherapy followed by concurrent chemoradiotherapy in locally advanced nasopharyngeal carcinoma patients whose EBV DNA remained detectable after one cycle neoadjuvant chemotherapy using GP regimen. The main question it aims to answer is: whether the addition of carrilizumab or nituzumab improve the treatment outcomes in the relatively poor prognostic patients identified by the response of EBV DNA. Participants will be randomized to the combination of carrilizumab and standard treatment , the combination of nituzumab and standard treatment or the standard treatment alone if their EBV DNA didn't decrease to undetectable level post first cycle of neoadjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly histologically confirmed non-keratinizing nasopharyngeal carcinoma, type of WHO II or III, EGFR+.
2. Age 18-70 years.
3. Clinical stage III-IVa (based on the 8th American Joint Committee on Cancer[AJCC] edition).
4. Patients with detectable pre-treatment plasma EBV DNA which remained detectable after one cycle neoadjuvant.
5. ECOG (Eastern Cooperative Oncology Group) score: 0-1
6. Hemoglobin (HGB) ≥90 g/L, white blood cell (WBC) ≥4×109 /L, platelet (PLT) ≥100×109 /L.
7. Liver function: Alanine transaminase(ALT), Aspartate aminotransferase(AST)< 1.5 times the upper limit of normal value (ULN), total bilirubin <1.0×ULN.
8. Renal function: serum creatinine <1×ULN.
9. Patients must sign informed consent and be willing and able to comply with the requirements of visits, treatment, laboratory tests and other research requirements stipulated in the research schedule.

Exclusion Criteria:

1. Histologically confirmed keratinizing squamous cell carcinoma (WHO I)
2. Suffered from other malignant tumors (except the cure of basal cell carcinoma or uterine cervical carcinoma in situ) previously.
3. Receiving radiotherapy or chemotherapy or targeted therapy previously
4. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant.
5. Patients with significantly lower heart, liver, lung, kidney and bone marrow function.
6. Severe, uncontrolled medical conditions and infections.
7. At the same time using other test drugs or in other clinical trials.
8. Refusal or inability to sign informed consent to participate in the trial.
9. Emotional disturbance or mental

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 459 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 3 years
  Defined from date of randomization to date of first documentation of progression or death due to any cause

SECONDARY OUTCOMES:
Overall survival | 3 years
  Defined from date of randomization to date of first documentation of death from any cause or censored at the date of the last follow-up.
Toxicities | 3 years
  Analysis of acute and late adverse events (AEs) are evaluated. Numbers of patients of treatment-related adverse events(acute toxicity) as assessed by CTCAE v5.0.Numbers of patients of late radiation toxicities were assessed using the Radiation Therapy Oncology Group and European Organization for Research and Treatment of Cancer late radiation morbidity scoring scheme.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan Universtiy Shanghai Cancer Centre, Shanghai, Shanghai Municipality, China